CLINICAL TRIAL: NCT03755050
Title: A 13-years Nationwide Retrospective Observational Study of Alpine Accidents in Austria - Sleighing, Skiing, Snowboarding, Snowshoeing, Climbing, Hiking, Cycling, Mountain Biking, Canyoning and Alpine Watersport Activities
Brief Title: A 13-years Nationwide Study of Alpine Accidents in Austria
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: AN2016-0018 358/4.8 390/5.5
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Alpine Accident; Sleighing; Climbing; Cycling; Canyoning; Hiking; Snowshoeing; Alpine Water-sport; Skiing/Snowboarding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Sleigh Accident: Accident while using a sleigh
  Interventions: Other: general and specific data
- Climbing Accident: Accident occurred while climbing (rock, ice)
  Interventions: Other: general and specific data
- Cycle Accident: Accident occurred while using any form of cycle in the mountains (e.g. bike, mountainbike, e-bike)
  Interventions: Other: general and specific data
- Canyoning Accident: Accident occurred while doing canyoning
  Interventions: Other: general and specific data
- Hiking Accident: Accident occurred while hiking in mountainous area.
  Interventions: Other: general and specific data
- Snowshoeing Accident: Accident occurred while doing Snowshoeing
  Interventions: Other: general and specific data
- Mountainous Water-sport Accident: Accident occurred while doing any type of Water-sport (e.g. canoeing, kayaking, tubing, swimming) in mountainous environment.
  Interventions: Other: general and specific data
- Skiing/Snowboarding: Accident occurred while using ski or a snowboard either in backcountry or on ski slope
  Interventions: Other: general and specific data

INTERVENTIONS:
Other: general and specific data — General and specific data collected

SUMMARY:
Brief Summary:

This observational study intends to analyze the characteristic of specific accidents happened in Austrian's mountainous regions. The mechanisms of accidents which are evaluated are accidents while using a sleigh, climbing accidents, cycle accidents, canyoning accidents, hiking accidents, snowshoeing accidents, water-sport accidents, ski and snowboard accidents.

DETAILED DESCRIPTION:
The data are collected retrospectively from the database of Austrian alpine police force. These data are analyzed. The information from this database (scene of accident, weather, daytime…) is compared to secondary data collected from the University Hospital of Innsbruck. The comparison of both databases was approved by the Austrian Data Protection Agency. The goal of the study is to give detailed information of circumstances leading to accident and give medical information of the patient's condition and his outcome.

The method to collect data and to analyze is the same than in AN4757 315/4.4 (NCT03405467).

ELIGIBILITY:
Inclusion Criteria:

* All patients with the criteria for an alpine accident characteristics described under "Conditions".

Exclusion Criteria:

* All patients without accident characteristics described under "Conditions".
* All patients which suffered an accident not in alpine environment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Patients in the two databases eligible for the searched injury patterns.
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2018-12-22 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of persons suffered an accident in Alpine Mountains in Austria | 2005-2018
  The number of persons which suffered one of the specified accidents. (n/year)
Gender of persons suffered an accident in Alpine Mountains in Austria | 2005-2018
  Gender male/female or non specified which suffered one of the specified accidents. (n/year)
Mortality of persons suffered an accident in Alpine Mountains in Austria | 2005-2018
  Number of persons deceased (deceased/n per year) which suffered one of the specified accidents.

SECONDARY OUTCOMES:
Number of patients treated per injury pattern at Medical University of Innsbruck, a major trauma center in western Austria. | 2005-2018
  (n/year) treated at Medical University of Innsbruck
Gender of patients treated per injury pattern at Medical University of Innsbruck, a major trauma center in western Austria. | 2005-2018
  male/female, unspecified treated at Medical University of Innsbruck (n/year)
Injury severity score (ISS) per injury pattern at Medical University of Innsbruck, a major trauma center in western Austria. | 2005-2018
  Injury severity score of suffered injury (ISS=AIS*AIS)
Abbreviated Injury severity scale (AIS) per injury pattern at Medical University of Innsbruck, a major trauma center in western Austria. | 2005-2018
  Abbreviated Injury Severity Scale of suffered injury (1-6 points; scale - minor, moderate, serious, severe, critical, maximum)
Type of evacuation | 2005-2018
  Type of evacuation (terrestrial, helicopter, combined terrestrial and helicopter) (n/year)
Mortality depending on evacuation type | 2005-2018
  Number of fatalities depending on type of evacuation (n/year)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ströhle, Principal Investigator — General and Surgical Critical Care Medicine, Medical University of Innsbruck
Locations (1):
- General and Surgical Critical Care Medicine, Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rugg CD, Malzacher T, Ausserer J, Rederlechner A, Paal P, Strohle M. Gender differences in snowboarding accidents in Austria: a 2005-2018 registry analysis. BMJ Open. 2021 Oct 19;11(10):e053413. doi: 10.1136/bmjopen-2021-053413. PMID 34667014